CLINICAL TRIAL: NCT03729986
Title: Activation Patterns of Respiratory Muscles to Loaded Inspiratory Muscle Tests in Healthy Adults Under Different Posture
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807021RINA
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-11

CONDITIONS: Accessory Muscle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy subjects without exercise habit that can cooperate with the measurements of this study, loaded inspiratory muscle test.
  Interventions: Other: Loaded inspiratory muscle test

INTERVENTIONS:
Other: Loaded inspiratory muscle test — Loaded inspiratory muscle tests will be set at 30% of maximal inspiratory pressure in sitting and supine positions. The orders of the two loaded test conditions will be conducted in random order with at least 20 minute separation. This is an observational study. Subjects will perform only 15 breaths with each loaded test condition to exam the performance of their inspiratory muscles. Loaded inspiratory muscle test is not for training.

SUMMARY:
Whether minimizing sternocleidomastoid (SCM) activation in supine position would increase diaphragm activation during loaded inspiratory muscle tests remains to be determined. Therefore, the purpose is to exam diaphragm and SCM activation during loaded inspiratory muscle tests in sitting and supine position in healthy adults.

DETAILED DESCRIPTION:
Inspiratory muscle training usually performed in the upright sitting position. In healthy individuals, sternocleidomastoid (SCM) is rarely recruited during tidal breathing, but previous studies have demonstrated SCM activation during loaded inspiratory muscle tests in upright sitting position. Whether minimizing SCM activation in supine position would increase diaphragm activation during loaded inspiratory muscle tests remains to be determined. Therefore, the purpose is to exam diaphragm and SCM activation during loaded inspiratory muscle tests in sitting and supine position in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years old
* without exercise habit (any exercise that less than 3 days/week)
* can cooperate with the measurements of this study

Exclusion Criteria:

* any clinical diagnosis that will influence the measurement, including any history of neuromyopathy
* angina, acute myocardial infarction in the previous one month
* pregnancy
* participated in inspiratory muscle training program in the previous three months
* any psychiatric or cognitive disorders, for example: Mini-Mental State Examination (MMSE) < 24, that will disturb the communication and cooperation of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults that are willing to cooperate the measurement of this study.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Diaphragm and Sternocleidomastoid muscle activation | Through the completion of the loaded inspiratory muscle test condition; it would take about 3 minutes
  Root mean square values during different conditions
The mean median frequency of diaphragm and sternocleidomastoid muscle | In one minute after the completion of the loaded inspiratory muscle test condition
  The power spectrum is divided into two equal areas of the frequency value by median frequency to exam muscle fatigability

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, Phd, Study Chair — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy of National Taiwan University, Taipei, Zhongzheng Dist, Taiwan